CLINICAL TRIAL: NCT02625311
Title: A Prospective Comparative Randomized International Multicenter Study Comparing MIS Computer Navigated Total Knee Arthroplasty vs Conventional Computer Navigated Total Knee Arthroplasty
Brief Title: Comparing Minimal Invasive Surgery en Conventional Total Knee Arthroplasty
Acronym: MIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC04-105
Record Dates: First submitted 2015-11-30; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — threonyl-lysyl-proline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIS (Experimental): Minimal invasive surgery for placement total knee prosthesis
  Interventions: Procedure: surgery method using CR TKP
- conventional approach (Active Comparator): conventional "open" surgery for placement total knee prosthesis.
  Interventions: Procedure: surgery method using CR TKP

INTERVENTIONS:
Procedure: surgery method using CR TKP — Operation through minimal invasive surgery or standard open surgery
  Other Names: Cruciate retaining (CR total knee prosthesis (TKP) Stryker

SUMMARY:
Randomized clinical trial comparing minimal invasive operating technique to conventional operating technique for placement of total knee prosthesis.

Clinical evaluations, patient questionnaires, X-rays and CT scans were done to compare these two techniques.

DETAILED DESCRIPTION:
Study executed with 3 centers and 69 patients.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring Total Knee Arthroplasty (TKA)
* patients with Osteo arthritis
* intact collateral ligaments and patella tendon
* patients willing and able to comply with the post-operative schedule

Exclusion Criteria:

* patients who require a revision TKA
* patients with TKA contralateral knee within 6 months with bad outcomes
* patients who need a TKA on contralateral side within 2 years
* intraoperative resurfacing of patella
* intraoperative eversion of patella
* patients who had prior procedure of involved knee such as high tibial osteotomy, cruciate ligament recontruction, knee fusion or patellectomy
* BMI > 30
* patients with fixed flexion contracture> 15 degrees
* patients with deformity greater than 20 degrees of varus or 15 degrees of valgus
* Patient with Mediolateral stability > 10 degrees patient with active or suspected malignancy
* patient with Rheumatoid arthritis
* patient with systemic disease that would effect subject's wellfare or overall outcome of the study
* patient with other severe concurrent joint involvement which can effect their outcome
* patients with an immobile hip
* patient with a history of Pulmonary embolism or Deep venous thrombosis

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-12; Primary Completion 2011-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
range of motion | pre-op vs post-op until 5 years post-op
  measurement of flexion and extension in degrees
blood loss | 24 hours after surgery
  measurement of milliliters blood loss during the first 24 hours after surgery

SECONDARY OUTCOMES:
patient questionnaire | pre-op vs post-op until 5 year post operative
  WOMAC pain and function score
chair rise and stair climb test | pre-op vs post-op until 5 years post operative
  Ability of patient rise from chair and climb stairs, amount of pain on VAS 1-10 does the patient have during these activities

REFERENCES:
- [Derived] Feczko P, Engelmann L, Arts JJ, Campbell D. Computer-assisted total knee arthroplasty using mini midvastus or medial parapatellar approach technique: A prospective, randomized, international multicentre trial. BMC Musculoskelet Disord. 2016 Jan 13;17:19. doi: 10.1186/s12891-016-0872-7. PMID 26762175